CLINICAL TRIAL: NCT02770183
Title: Rate of Left Ventricular Systolic Function's Recuperation After Cardiac Surgery With Extracorporeal Circulation.
Acronym: Imacor-1
Status: Withdrawn | Type: Observational
Why Stopped: Problems with grant
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Samuele Ceruti, MD, University Hospital, Geneva
Other Study IDs: CERU-1601
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Stunning; Transesophageal Echocardiography; Circulation, Extracorporeal
Keywords: Myocardial stunning; Echocardiography, Transesophageal; Extracorporeal Circulation
MeSH Terms: conditions — Myocardial Stunning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive patients: Consecutive patients waiting to have elective cardiac surgery will be eligible. Each week the principal investigator will track patients in the operating program. The day of the consultation or the day before the operation, one of the investigators will have a talk with the patient to provide information and clarify doubts, also allowing the patient to read and look good all the details before giving its approval. For the screening, the principal investigator will use the criteria of inclusion and exclusion to select patients for the study. The screening uses clinical, laboratory or without other biological information.
  To minimize confounding factors, it will be taken consecutive patients, that will also be analyzed regarding all known variables that can affect the systolic function, as non-modifiable (age, cardiovascular risk factors, heart-rate variability and preoperative basal systolic function) and modifiable.
  Interventions: Device: Imacor

INTERVENTIONS:
Device: Imacor — In ICU, the doctors in charge places the probe in the esophagus, executing a series of morphological evaluations and semi-quantitative evaluations. Each image is saved as a video loop or a static image, to have a basic data for each patient and perform an off-line analysis. At the end of the first recording, the esophageal probe is left in the neutral position in the stomach, to eliminate any risk associated with a local increase of pressure.
  During the stay in the intensive care unit until the end of the study, the esophageal probe will be left in the neutral position, to run every two hours a new echocardiographic assessment on the main window, similar to the first evaluation, always recording loop-video and photographs, to have a time course of recovery of cardiac contractile function. All images will be stored in a digital archive.
  Other Names: hTEE

SUMMARY:
The rational of the study is the description of the evolution of systolic cardiac function post-stunning, evaluated by transesophageal minimally invasive echocardiography (hTEE). The uses of these non-invasive methods have proved to be accurate for the qualitative and semi-quantitative determination of the contractile function of the left ventricle and the volume status of the patient. Furthermore the use of this technique has been demonstrated to be a reliable method to analyze the stunning recovery infarction after controlled cardiac arrest during the extra-corporeal circulation.

DETAILED DESCRIPTION:
Myocardial stunning is a secondary pathophysiologic condition for a sustained reduction in myocardial perfusion, which produces kinetic abnormalities in left ventricular wall that persist for hours or days after the reperfusion phase. The physiological elements of the stunning are: a) reduction in coronary blood flow, b) a partial or complete restoration of coronary artery circulation and c) the dysfunction of persistence for a limited period, but longer compared to recovery coronaire's flow.

Cardiac surgery with cardiopulmonary bypass is a leading cause of bewilderment myocardique. This technique associated with administering a cardioplegic solution used to stop the heart and myocardial protection on ischemia see myocardique consideration. It typically also secondary to secondary inflammatory condition in the extracorporeal circulation and the ischemia-reperfusion phenomenon (formation of free radicals), also with the important activation coagulation. Myocardial stunning occurs in suites aortic unclamping during cardiopulmonary bypass. Cold ischemia performed by a cardioplegic liquid at 4 °C results in reduced energy demands and thus to maintain some balance between metabolism, perfusion and myocardial function during coronary by-pass. When aortic unclamping, there is usually a pure myocardial stunning (without necrosis). After the coronary by-pass, the myocardial thickening fraction is unchanged in the immediate future, but significantly decreased in the hours before a full recovery between the following hours. In the factors associated with changes in systolic function, autonomic nervous system is responsible for the regulation of blood pressure and heart function in response to the stress of the coronary by-pass and the postoperative state. Reduced variability in heart rate (heart rate variability - HRV) heard how sign of autonomic dysfunction is also associated with myocardial stunning with a rate of cardiaque post-surgery complications high.

So far no group has had the opportunity to study "in vivo" the temporal evolution of myocardial stunning after the coronary by-pass as an example of myocardial stunning "controlled" in order to better understand the pathophysiology of 'event. Indeed, the basis of myocardial function recovery time following coronary by-pass is unknown and the impact of intraoperative procedures on this recovery.

Transesophageal echocardiography, that is the gold standard for assessment of systolic function, has gradually gained popularity and is used daily in the ICU to evaluate the patient's hemodynamic status and evaluation of contractile function of the left ventricle to load. One of its advantages is to measure heart activity at the bedside and assist the physician in intensive care in the management of hemodynamic acute changes. It also allows also to analyze the response to treatment defined above. Among the limitations of transesophageal echocardiography are: the need for intensivists to be relevant to this technique, the discontinuous nature of the procedure ( "one shot" monitoring) and finally semi-invasif character that make it difficult 'prolonged and repeated execution of the various measures.

Recent improvement in electronics has enabled the development of miniaturized sensors for hemodynamic transesophageal echocardiography (ImaCor® ClariTEE®), called hTEE (hemodynamic trans-esophageal echocardiography), which are used to perform an extended hemodynamic monitoring ventilated patients; these prototypes are not yet widespread in Intensive Care Unit; their diagnostic capabilities and therapeutic impacts are currently under clinical research. been studies in the past allowed us to validate the clinical image quality and how the clinical information obtained are useful for clinical management of patient. In particular, these studies have demonstrated the ease with which thanks to the small size of the probe, the feedback of the superior vena cava, the patient's volume status, left ventricular systolic function based on the Fractional Area Change, the size of the right ventricle, and a pericardial effusion and cardiac tamponade during the first test of positioning sonde.

The advantages of continuous Htee of this new technique are related to the small size of the probe, ease of positioning the probe in the esophagus, the diagnostic reliability and the ability to stay up to 72 hours because the risk of pressure sores or lesions are comparable to those of a nasogastric feeding tube (which is the same size). Compared to the conventional trans-esophageal echocardiography, hTEE offers the advantage of performing continuous monitoring rather than a case-by case basis. In particular, for the study of post-operative myocardial stunning, this technique allows for a verification of the time course of myocardial stunning, and thus describe the pathophysiology and the kinetics of recovery of left ventricular contractile function. Furthermore this technique provides the means to identify perioperative factors that can change this recovery (induce or shorten).

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years), waiting for a heart surgery
* Patients of both sexes
* Patients hospitalized in intensive care after the operation
* Informed consent available

Exclusion Criteria:

* Patients with contraindications to the placement of a nasogastric tube for the presence of esophageal varices, esophageal lesions or esophageal-gastric complications known.
* Patients with severe sepsis or septic shock, according to international definitions.
* Patients with severe coagulopathy defined as a lower thrombocytopenia at 20 G / L and / or INR> 2.5 and / or aPTT in the therapeutic range and / or an anti-Xa activity in the ultra-therapeutic range and / or a fibrinogen value less than 1 g / L.
* Patients with poor prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients waiting to have elective cardiac surgery needing a cardiopulmonary by-pass will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fractional Area Change analysis | 72 hours
  Primary outcome is the evolution of Fractional Area Change for the duration of the study. The assessment of cardiac contractile function, which method is better described below, will be based mainly on a serial analysis of the Fractional Area Change and semi-quantitative assessment of ejection fraction in projection 4 cavities.

SECONDARY OUTCOMES:
Stratify patients | 72 hours
  Identify the presence of specific subgroups of patients, that will correlate the recovery rate of the systolic function with all other clinical, demographic and operational variables, as biologic parameters (age, sex), clinical parameters (like preoperative disease, use of B-blockers, preoperative left-ventricular-ejection-fraction, any dysfunction of sinoatrial node or the recovery of heart rate variability) and peri-operative parameters (like duration of extra-corporeal circulation, type of cardioplegia, duration of surgery, use of amine, hemoglobin values after surgery, etc...)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Bendjelid, Prof., Study Director — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heyndrickx GR, Millard RW, McRitchie RJ, Maroko PR, Vatner SF. Regional myocardial functional and electrophysiological alterations after brief coronary artery occlusion in conscious dogs. J Clin Invest. 1975 Oct;56(4):978-85. doi: 10.1172/JCI108178. PMID 1159098
- [Result] Braunwald E, Kloner RA. The stunned myocardium: prolonged, postischemic ventricular dysfunction. Circulation. 1982 Dec;66(6):1146-9. doi: 10.1161/01.cir.66.6.1146. PMID 6754130
- [Result] Marban E. Myocardial stunning and hibernation. The physiology behind the colloquialisms. Circulation. 1991 Feb;83(2):681-8. doi: 10.1161/01.cir.83.2.681. No abstract available. PMID 1991384
- [Result] Bolli R. Myocardial 'stunning' in man. Circulation. 1992 Dec;86(6):1671-91. doi: 10.1161/01.cir.86.6.1671. No abstract available. PMID 1451239
- [Result] Warren OJ, Watret AL, de Wit KL, Alexiou C, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 2--anti-inflammatory therapeutic strategies. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):384-93. doi: 10.1053/j.jvca.2008.09.007. Epub 2008 Dec 3. No abstract available. PMID 19054695
- [Result] Wan S, LeClerc JL, Vincent JL. Inflammatory response to cardiopulmonary bypass: mechanisms involved and possible therapeutic strategies. Chest. 1997 Sep;112(3):676-92. doi: 10.1378/chest.112.3.676. PMID 9315800
- [Result] Day JR, Taylor KM. The systemic inflammatory response syndrome and cardiopulmonary bypass. Int J Surg. 2005;3(2):129-40. doi: 10.1016/j.ijsu.2005.04.002. Epub 2005 Aug 1. PMID 17462274
- [Result] Dixon B, Santamaria J, Campbell D. Coagulation activation and organ dysfunction following cardiac surgery. Chest. 2005 Jul;128(1):229-36. doi: 10.1378/chest.128.1.229. PMID 16002940
- [Result] Esmon CT. The interactions between inflammation and coagulation. Br J Haematol. 2005 Nov;131(4):417-30. doi: 10.1111/j.1365-2141.2005.05753.x. PMID 16281932
- [Result] Compostella L, Russo N, Compostella C, Setzu T, D'Onofrio A, Isabella G, Tarantini G, Iliceto S, Gerosa G, Bellotto F. Impact of type of intervention for aortic valve replacement on heart rate variability. Int J Cardiol. 2015 Oct 15;197:11-5. doi: 10.1016/j.ijcard.2015.06.004. Epub 2015 Jun 14. PMID 26113470
- [Result] Vieillard-Baron A, Prin S, Chergui K, Dubourg O, Jardin F. Hemodynamic instability in sepsis: bedside assessment by Doppler echocardiography. Am J Respir Crit Care Med. 2003 Dec 1;168(11):1270-6. doi: 10.1164/rccm.200306-816CC. No abstract available. PMID 14644922
- [Result] Etchecopar-Chevreuil C, Francois B, Clavel M, Pichon N, Gastinne H, Vignon P. Cardiac morphological and functional changes during early septic shock: a transesophageal echocardiographic study. Intensive Care Med. 2008 Feb;34(2):250-6. doi: 10.1007/s00134-007-0929-z. Epub 2007 Nov 15. PMID 18004543
- [Result] Vignon P, Mentec H, Terre S, Gastinne H, Gueret P, Lemaire F. Diagnostic accuracy and therapeutic impact of transthoracic and transesophageal echocardiography in mechanically ventilated patients in the ICU. Chest. 1994 Dec;106(6):1829-34. doi: 10.1378/chest.106.6.1829. PMID 7988209
- [Result] Slama MA, Novara A, Van de Putte P, Diebold B, Safavian A, Safar M, Ossart M, Fagon JY. Diagnostic and therapeutic implications of transesophageal echocardiography in medical ICU patients with unexplained shock, hypoxemia, or suspected endocarditis. Intensive Care Med. 1996 Sep;22(9):916-22. doi: 10.1007/BF02044116. PMID 8905426
- [Result] Vieillard-Baron A, Slama M, Mayo P, Charron C, Amiel JB, Esterez C, Leleu F, Repesse X, Vignon P. A pilot study on safety and clinical utility of a single-use 72-hour indwelling transesophageal echocardiography probe. Intensive Care Med. 2013 Apr;39(4):629-35. doi: 10.1007/s00134-012-2797-4. Epub 2013 Jan 4. PMID 23287876
- [Result] Treskatsch S, Balzer F, Knebel F, Habicher M, Braun JP, Kastrup M, Grubitzsch H, Wernecke KD, Spies C, Sander M. Feasibility and influence of hTEE monitoring on postoperative management in cardiac surgery patients. Int J Cardiovasc Imaging. 2015 Oct;31(7):1327-35. doi: 10.1007/s10554-015-0689-8. Epub 2015 Jun 6. PMID 26047772
- [Result] Begot E, Dalmay F, Etchecopar C, Clavel M, Pichon N, Francois B, Lang R, Vignon P. Hemodynamic assessment of ventilated ICU patients with cardiorespiratory failure using a miniaturized multiplane transesophageal echocardiography probe. Intensive Care Med. 2015 Nov;41(11):1886-94. doi: 10.1007/s00134-015-3998-4. Epub 2015 Aug 8. PMID 26254013
- [Result] Imren Y, Tasoglu I, Oktar GL, Benson A, Naseem T, Cheema FH, Unal Y. The importance of transesophageal echocardiography in diagnosis of pericardial tamponade after cardiac surgery. J Card Surg. 2008 Sep-Oct;23(5):450-3. doi: 10.1111/j.1540-8191.2008.00581.x. Epub 2008 May 7. PMID 18462344